CLINICAL TRIAL: NCT06455059
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of Vosoritide in Children With Hypochondroplasia
Brief Title: Interventional Study of Vosoritide for the Treatment of Children With Hypochondroplasia
Acronym: CANOPY-HCH-3
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 111-303
Record Dates: First submitted 2024-06-07; First posted 2024-06-12 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Hypochondroplasia
Keywords: Hypochondroplasia; Dwarfism; Bone Diseases; Bone Disease, Developmental; HCH; Natriuretic Peptide, C-Type; Musculoskeletal Diseases; Natriuretic Agents; Physiological Effects of Drugs; Skeletal Dysplasias; Genetic Diseases, Inborn; Osteochondrodysplasias; Vosoritide; Voxzogo
MeSH Terms: conditions — Hypochondroplasia; Dwarfism; Bone Diseases; Bone Diseases, Developmental; Musculoskeletal Diseases; Genetic Diseases, Inborn; Osteochondrodysplasias | interventions — vosoritide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vosoritide injection with vial and syringe (Experimental)
  Interventions: Drug: Vosoritide
- Placebo injection with vial and syringe (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Vosoritide — Subcutaneous injection of recommended dose of vosoritide based on weight-band dosing once daily.
  Other Names: Modified recombinant human C-type natriuretic peptide
  Arms: vosoritide injection with vial and syringe
Drug: Placebo — Subcutaneous injection of recommended dose of placebo
  Arms: Placebo injection with vial and syringe

SUMMARY:
The intent and design of this Phase 3 study is to assess vosoritide as a therapeutic option for the treatment of children with hypochondroplasia (HCH).

DETAILED DESCRIPTION:
This is a Phase 3 randomized, stratified, placebo-controlled, double-blind multicenter study to evaluate the effect of 52 weeks of daily vosoritide administration on annualized growth velocity (AGV) in participants with HCH. Eligible participants with documented HCH confirmed by genetic testing will roll over from Study 111-902 and enter the 111-303 study. Participants will be randomly assigned to one of two treatment groups: Placebo or Vosoritide. The route of administration is subcutaneous injection, and the frequency of administration is daily.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must be ≥ 3 to < 18 years of age at enrollment
2. A confirmed genetic diagnosis of HCH
3. A height Z score of ≤ - 2.0 standard deviations (SDs) in reference to the general population of the same age and sex, as calculated using the Center for Disease Control and Prevention (CDC) growth charts
4. Males and females are eligible to participate in this clinical study.
5. Females ≥ 10 years old or who have begun menses must have a negative pregnancy test at the Screening Visit and be willing to have additional pregnancy tests during the study.
6. If sexually active, participants must be willing to use a highly effective method of contraception while participating in the study.

Exclusion Criteria:

1. Short stature condition other than HCH
2. Have an unstable condition likely to require surgical intervention during the study.
3. Evidence of decreased growth velocity and/or growth plate closure
4. Taking any of the prohibited medications
5. Treated with growth hormone, insulin-like growth factor 1 (IGF-1), or anabolic steroids
6. Planned or expected to have limb-lengthening surgery during the study period.
7. Planned or expected bone-related surgery (ie, surgery involving disruption of bone cortex, excluding tooth extraction), during the study period
8. Require any investigational agent prior to completion of study period.
9. Received vosoritide or another investigational product or investigational medical device in the past
10. Have used any investigational product or investigational medical device for the treatment of HCH or short stature at any time, including vosoritide
11. Have current malignancy, history of malignancy, or currently under work-up for suspected malignancy.
12. Have known hypersensitivity to vosoritide or its excipients.
13. Concurrent disease or condition that, in the view of the investigator, would interfere with study participation or safety evaluations, for any reason.

Ages: 3 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in annualized growth velocity (AGV) at Week 52 versus placebo | At week 52

SECONDARY OUTCOMES:
Change from baseline in standing height at Week 52 versus placebo | At week 52
Change from baseline in height Z-score at Week 52 versus placebo | At week 52

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — BioMarin Pharmaceutical
Locations (23):
- United States (4):
  - Nemours Alfred I. DuPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Murdoch Children's Research Institute, Parkville, Victoria, Australia
- Canada (3):
  - University of Alberta Stollery Children's Hospital, Edmonton, Alberta
  - SickKids - The Hospital for Sick Children, Toronto, Ontario
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal, Quebec
- France (4):
  - Hospices Civils de Lyon - Hopital Femme Mere Enfant, Lyon
  - Hopital de la Timone, Marseille
  - Hopital Necker-Enfants Malade, Paris
  - CHU de Toulouse, Toulouse
- Germany (2):
  - Uniklinik Koln, Cologne
  - Univeristatskinderklinik Magdeburg, Magdeburg
- Italy (3):
  - Instituto Giannina Gaslini, Genoa
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome
  - Ospedale Pediatrico Bambino Gesu, Rome
- Japan (4):
  - Osaka University Hosptial, Osaka
  - Tokushima University Hospital, Tokushima
  - Institute of Science Tokyo Hospital, Tokyo
  - Tottori University Hospital, Tottori
- Vithas Hospital San Jose, Vitoria-Gasteiz, Spain
- Great Ormond Street Hospital for Children NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No